CLINICAL TRIAL: NCT04309929
Title: Description of the Analgesia Obtained With the Anesthesiological Protocols Currently Used in Breast Surgery
Status: Completed | Type: Observational
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Villa, Principal investigator, Careggi Hospital
Other Study IDs: CEAVC OSS. 16.246
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Cancer; Breast; Mastectomy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Analgesics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with breast cancer: Female patients (age> 18yrs) in ASA class <4; candidate for a planned surgery for simple mastectomy, simple mastectomy with immediate reconstruction, mastectomy with sentinel node biopsy, modified radical mastectomy (unilateral or bilateral)
  Interventions: Drug: Analgesics

INTERVENTIONS:
Drug: Analgesics — All patients will undergo the anesthesiological and surgical treatment provided for the patient's clinical conditions and in no case will the patients undergo a change in the normal diagnostic-therapeutic path due to participation in this study.

SUMMARY:
This study aims to describe the pain-relieving effect obtained with the current post-surgery pain control methods used in breast surgery by measuring the painful sensation and the consumption of opioids in the first 24 post-surgery hours. It also aims to describe the appearance of any complications such as post-surgery nausea and vomiting. Current anesthesia involves the combined use of intravenous painkillers and anti-inflammatory drugs such as acetaminophen, ketorolac, tramadol or morphine (the latter via PCA system = patient-controlled analgesia) or for local administration at the surgical site level ( local anesthetics). It is also proposed to describe the intensity and interference of pain in daily activities

DETAILED DESCRIPTION:
Breast cancer is the second most common in the world and the most frequent in the female population. In Italy, around 48,000 new cases were diagnosed in 2013. Every year patients undergoing surgical procedures in the region of the breast and armpit, like other surgical areas, report a significant incidence of acute postoperative pain which in 25-60% of cases can progress to chronic pain and therefore it needs a timely and effective control.

Breast surgery is associated with a high incidence of postoperative nausea and vomiting (PONV) whose etiology is multifactorial and includes factors such as age, type of intervention, positive history of PONV and, primarily, the amount of morphine used to ensure postoperative analgesia, the type of anesthesia and the intensity of postoperative pain.

The conventional anesthesiological approach to breast surgery involves the use of general anesthesia and postoperative analgesic therapy based on opiates and fans. Some techniques of locoregional anesthesia such as paravertebral block, thoracic peridural analgesia and intercostal block, associated with sedoanalgesia or general anesthesia, have joined the standard anesthesiological conduct helping to improve pain control, response to surgical stress, post-operative respiratory function, the incidence of thromboembolic events and it seems they can also contribute to reducing the incidence of distant metastases. In addition, making possible a reduced use of opiates further decrease the incidence of PONV. As part of this multimodal approach to anesthesia and analgesia for breast surgery, PECS Block I and II and the Serratus Plane Block (SPB) have recently been introduced into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age> 18 years;
* Patients in ASA class <4;
* Planned mastectomy surgery, simple mastectomy with immediate reconstruction, mastectomy with sentinel-lymph node biopsy, modified radical mastectomy (unilateral or bilateral);
* Absence of allergies or hypersensitivity reported and / or documented to drugs used routinely for post-operative analgesia;
* Absence of inflammatory changes at the surgical site level;
* Presence of the patient's informed consent to the processing of personal data;

Exclusion Criteria:

* Known alterations of coagulation;
* Known cardiac arrhythmias (atrial sinus block I, II, III type, atrioventricular block I, II and III type);
* Documented renal failure (patient undergoing renal replacement therapy, or creatininemia ≥ 2 mg / dl);
* Severe hepatic insufficiency (Child-Plugh class III and IV); Seizure states (absences, seizures of large and / or small epileptic disease);
* Respiratory failure (PaO2 ≤ 60mmHg PaCO2≥ 50mmHg);

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who in accordance with the inclusion and exclusion criteria have given their consent to the processing of personal data will be considered for analysis. All patients will undergo the anesthesiological and surgical treatment foreseen for the patient's clinical condition and in no case will the patients undergo a modification of the normal diagnostic-therapeutic path due to participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the change of level of anesthesia | Up to 24 hours after surgery
  Describing the level of analgesia obtained in the first 24 hours post-operative in patients undergoing simple mastectomy, mastectomy with immediate reconstruction with expander or retropectoral prosthesis, mastectomy with sentinel node biopsy and radical mastectomy modified with the anesthesiological protocols used routinariamentally. Analgesia will be evaluated every 6 hours and for the first 24 post-operative hours (at 0, 6, 12, 18, 24 hours from the end of the surgical intervention) through the NRS (Numerical Rating Scale).
  The Numerical Rating Scale is a pain sensation rating scale at points where the patient chooses a value ranging from 0 (no pain) to 10 (maximum pain). From 1 to 3 it is considered mild pain, from 4-7 moderate, from 8-10 severe.

SECONDARY OUTCOMES:
Describing the total amount of morphine used in the first 24 post-operative hours. | 24 hours after surgery
  The total amount of morphine used will be expressed in milligrams of morphine used by the patient in the first 24 hours post-operative normalized per kilogram of body weight (mg / kg).
Describing the incidence of PONV (Postoperative Nausea and Vomiting). | 24 hours after surgery
  The incidence of PONV, measured at 0, 6, 12, 18 and 24 hours will be expressed in terms of percentage.
Describing of change in severity of PONV (Postoperative Nausea and Vomiting). | 24 hours after surgery
  The incidence of PONV, measured at 0, 6, 12, 18 and 24 hours will be expressed in terms of percentage. The severity of PONV will be expressed according to the following evaluation scheme: absence of nausea = 0, mild nausea = 1, moderate = 2, severe nausea or vomiting = 3
Description of the change of the intensity of pain on daily activities reported by patients undergoing breast surgery. | 3 months after surgery
  The painful sensation is assessed by six questions on the quality of pain experienced in the previous 24 hours; for each question, an answer corresponding to a numerical value from 0 (no pain) to 10 (maximum) according to the Numerical Rating Scale (NRS) is requested and recorded. In addition, the percentage of relief provided by analgesic drugs, possibly taken, is investigated by administering a question and recording a percentage value, from 0% (minimum) to 100% (maximum), referring to the percentage sensation of pain relief. A second question is requested related to the type of drug possibly taken. At the end of the questionnaire, an overall score is calculated regarding the questions on the intensity of pain (0-40, 0-10 points for each answer to questions 3 to 6). A score of 0 (no pain) to 10 (maximum pain) is referred to the percentage of relief given by the analgesics corresponding to the value given in percentage / 10.
Description of the change of the interference of pain on daily activities reported by patients undergoing breast surgery. | 3 months after surgery
  The interference of pain includes the evaluation of 7 fields referring to which patients can express for each field, according to a numerical scale from 0 (minimum) to 10 (maximum), how much pain interferes. The numerical scale from 0-10 allows to record a response that varies between 0 = no interference in the activity, and 10 = completely interferes with the activity. This scale has been validated according to psychometric criteria. At the end of the questionnaire, an overall score is calculated regarding the questions on the intensity of pain (0-40, 0-10 points for each answer to questions 3 to 6). A score from 0-10 refers to the percentage of relief given by the analgesics corresponding to the value given as a percentage / 10. An overall score is calculated from 0 (no interference) to 70 (maximum interference), from 0 to 10 for each of the seven fields.
Description of the change of the incidence and impact on daily activities of the pain reported by patients undergoing breast surgery. | 3 months after surgery
  The incidence on daily pain activities will be assessed 3 months after surgery through the Brief Pain Inventory (BPI ) scale in the Italian validated version. The Brief Pain Inventory questionnaire evaluates the multidimensional experience of pain through two domains: the intensity of pain and the interference of pain (see the following outcome) in daily activities.An overall final score is calculated from 0 (minimum) to 120 (maximum) corresponding to the multidimensional experience of pain, obtained from outcomes 5 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Guido, MD, Principal Investigator — Careggi Hospital
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

REFERENCES:
- [Background] Gewandter JS, Dworkin RH, Turk DC, Farrar JT, Fillingim RB, Gilron I, Markman JD, Oaklander AL, Polydefkis MJ, Raja SN, Robinson JP, Woolf CJ, Ziegler D, Ashburn MA, Burke LB, Cowan P, George SZ, Goli V, Graff OX, Iyengar S, Jay GW, Katz J, Kehlet H, Kitt RA, Kopecky EA, Malamut R, McDermott MP, Palmer P, Rappaport BA, Rauschkolb C, Steigerwald I, Tobias J, Walco GA. Research design considerations for chronic pain prevention clinical trials: IMMPACT recommendations. Pain. 2015 Jul;156(7):1184-1197. doi: 10.1097/j.pain.0000000000000191. PMID 25887465
- [Background] Kairaluoma PM, Bachmann MS, Korpinen AK, Rosenberg PH, Pere PJ. Single-injection paravertebral block before general anesthesia enhances analgesia after breast cancer surgery with and without associated lymph node biopsy. Anesth Analg. 2004 Dec;99(6):1837-1843. doi: 10.1213/01.ANE.0000136775.15566.87. PMID 15562083
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] AIRTUM Working Group. Italian cancer figures, report 2013: Multiple tumours. Epidemiol Prev. 2013 Jul-Oct;37(4-5 Suppl 1):1-152. English, Italian. PMID 24259384
- [Background] Katz J, Poleshuck EL, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for acute pain and its persistence following breast cancer surgery. Pain. 2005 Dec 15;119(1-3):16-25. doi: 10.1016/j.pain.2005.09.008. Epub 2005 Nov 17. PMID 16298063
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Lynch EP, Welch KJ, Carabuena JM, Eberlein TJ. Thoracic epidural anesthesia improves outcome after breast surgery. Ann Surg. 1995 Nov;222(5):663-9. doi: 10.1097/00000658-199511000-00009. PMID 7487214
- [Background] Aufforth R, Jain J, Morreale J, Baumgarten R, Falk J, Wesen C. Paravertebral blocks in breast cancer surgery: is there a difference in postoperative pain, nausea, and vomiting? Ann Surg Oncol. 2012 Feb;19(2):548-52. doi: 10.1245/s10434-011-1899-5. Epub 2011 Jul 16. PMID 21769470
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Bouzinac A, Tournier JJ, Merouani M, Delbos A. [Sensory blockade and efficiency of the "pec block 2" for postoperative analgesia after breast cancer surgery]. J Gynecol Obstet Biol Reprod (Paris). 2015 Jan;44(1):98-9. doi: 10.1016/j.jgyn.2014.09.004. Epub 2014 Oct 1. No abstract available. French. PMID 25282097
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Sopena-Zubiria LA, Fernandez-Mere LA, Valdes Arias C, Munoz Gonzalez F, Sanchez Asheras J, Ibanez Ernandez C. [Thoracic paravertebral block compared to thoracic paravertebral block plus pectoral nerve block in reconstructive breast surgery]. Rev Esp Anestesiol Reanim. 2012 Jan;59(1):12-7. doi: 10.1016/j.redar.2011.10.001. Epub 2012 Mar 14. Spanish. PMID 22429631
- [Background] Langford R, Brown I, Vickery J, Mitchell K, Pritchard C, Creanor S. Study protocol for a double blind, randomised, placebo-controlled trial of continuous subpectoral local anaesthetic infusion for pain and shoulder function following mastectomy: SUB-pectoral Local anaesthetic Infusion following MastEctomy (SUBLIME) study. BMJ Open. 2014 Sep 30;4(9):e006318. doi: 10.1136/bmjopen-2014-006318. PMID 25270861
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Derived] Villa G, Mandarano R, Scire-Calabrisotto C, Rizzelli V, Del Duca M, Montin DP, Paparella L, De Gaudio AR, Romagnoli S. Chronic pain after breast surgery: incidence, associated factors, and impact on quality of life, an observational prospective study. Perioper Med (Lond). 2021 Feb 24;10(1):6. doi: 10.1186/s13741-021-00176-6. PMID 33622393
- See also: Globocan 2012 — http://globocan.iarc.fr/Default.aspx